CLINICAL TRIAL: NCT02665975
Title: Internet-based Versus Face-to-face Clinical Care for Tinnitus: A Multi-study Randomised Control Trial
Brief Title: Internet-based Versus Face-to-face Clinical Care for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARU-0116
Record Dates: First submitted 2016-01-22; First posted 2016-01-28 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2019-07

CONDITIONS: Tinnitus
Keywords: Tinnitus treatment; Internet-intervention; CBT
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group: iCBT (Experimental): CBT-based internet-intervention for tinnitus The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8 week long e-learning intervention, with new modules introduced weekly and assignments given to practice techniques learnt.
  Interventions: Behavioral: CBT-based internet-intervention for tinnitus
- Face-to-face clinical tinnitus care (Active Comparator): Receive individual face-to-face tinnitus care, and follow-up appointments as required.
  Interventions: Behavioral: Face-to-face clinical tinnitus care

INTERVENTIONS:
Behavioral: CBT-based internet-intervention for tinnitus — Tinnitus e-learning programme
  Other Names: iCBT
  Arms: Experimental group: iCBT
Behavioral: Face-to-face clinical tinnitus care — Hospital tinnitus counselling
  Arms: Face-to-face clinical tinnitus care

SUMMARY:
The purpose of this study is to compare the effectiveness of a CBT-based internet intervention with face to face standard clinical care for adults with tinnitus in the United Kingdom.

DETAILED DESCRIPTION:
Objectives Tinnitus is one of the most distressing disabilities and innovative ways of managing the related health care burden is required. A cognitive behavioural therapy (CTB) based internet intervention (iCBT) has been developed to improve access to tinnitus treatments. This study aims to determine the feasibility and effectiveness of iCBT in reducing the impact associated with tinnitus in the United Kingdom (UK) compared to standard face-to-face clinical care.

Design A two-armed Randomized Control Trial (RCT), will be used to evaluate the effectiveness iCBT on tinnitus distress. Participants placed in the experimental group will receive iCBT and those in the control group will undergo standard face-to-face hospital based clinical care.

Setting: This will be an multi-center study, recruiting from three tinnitus clinics in the East of England, UK; namely: Norfolk and Norwich University Hospital Trust, Milton Keynes University Hospital and Hinchingbrooke Healthcare NHS Trust

Participants: Recruitment will be undertaken from 3 separate clinical settings. Adult patients seen by ENT Consultants or Audiologist at these centers who mention being significantly bothered by tinnitus, and who would normally be referred for tinnitus services will be considered for the study. 80 Participants will be recruited and will be randomly assigned to either receiving face-to-face clinical clinical care consisting or or internet-based intervention (iCBT).

Intervention:

i) iCBT group: This group will undergo a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8 week long e-learning intervention, with new modules introduced weekly and assignments given to practice techniques learnt.

ii) Standard clinical care group: receive individual face-to-face tinnitus appointment providing the care deemed most important to this individual and follow-up appointments as required.

Outcome measures: The main outcome measure is the Tinnitus Functional Index. Secondary outcome measures are the Tinnitus Handicap Inventory- Screening version and self-reported measures for insomnia, hearing disability, cognitive functioning, hyperacusis, anxiety and depression and quality of life. These will be measured at baseline, 3 months post- intervention and 6-months post- intervention, to assess the intervention effects over time.

Hypothesis: If iCBT proves feasible and is effective compared to standard clinical care, it may have implications for the way tinnitus suffers are managed in the UK. It may be that a subset of tinnitus suffers can be managed though an e-learning treatment program, freeing up services for those with more severe problems that need face to face treatment.

ELIGIBILITY:
Inclusion Criteria:

* Attending either Norfolk and Norwich University Hospital, Milton Keynes University Hospital or Hinchingbrooke Hospitals as recruitment is via these hospitals
* The ability to read and type in English
* No barriers to using a computer (e.g. significant fine motor control or visual problems)
* Internet and e-mail access, and the ability to use these
* Commitment to completing the programme
* Completion of the online screening and outcome questionnaires
* Agreeing to participate in either group and be randomized to one of these groups
* Understanding and working towards the end goal of reducing the impact and distress of tinnitus, although the strength of the tinnitus may remain the same

Exclusion Criteria:

* Reporting any major medical or psychiatric conditions
* Reporting pulsatile, objective or unilateral tinnitus, which have not been investigated medically
* Tinnitus as a consequence of a medical disorder, still under investigation
* Undergoing any tinnitus therapy concurrently to partaking in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Peter, Study Chair — Anglia Ruskin University
Locations (3):
- United Kingdom (3):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Hinchingbrooke Hospital, Huntingdon
  - Milton Keynes University Hospital, Milton Keynes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigo H, Beukes EW, Andersson G, Manchaiah V. Internet-based cognitive-behavioural therapy for tinnitus: secondary analysis to examine predictors of outcomes. BMJ Open. 2021 Aug 20;11(8):e049384. doi: 10.1136/bmjopen-2021-049384. PMID 34417217
- [Derived] Beukes EW, Andersson G, Allen PM, Manchaiah V, Baguley DM. Effectiveness of Guided Internet-Based Cognitive Behavioral Therapy vs Face-to-Face Clinical Care for Treatment of Tinnitus: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Dec 1;144(12):1126-1133. doi: 10.1001/jamaoto.2018.2238. PMID 30286238
- [Derived] Beukes EW, Baguley DM, Allen PM, Manchaiah V, Andersson G. Guided Internet-based versus face-to-face clinical care in the management of tinnitus: study protocol for a multi-centre randomised controlled trial. Trials. 2017 Apr 21;18(1):186. doi: 10.1186/s13063-017-1931-6. PMID 28431551

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Started | 46 | 46
Completed | 37 | 37
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Population: Both intention to treat and pre-protocol analysis used
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.65 (12.19) | 55.26 (11.62) | 52.96 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 29 | 26 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Tinnitus Functional Index Score at Baseline [Mean (Standard Deviation); unit: scores on a scale at baseline] — A measure of tinnitus severity. Measured on a scale of 0 to 100. Lower scores indicate less severe tinnitus. A score of 25 or higher indicates the need for an intervention. A score of 50 or above indicates severe tinnitus. If post-intervention scores are lower than baseline it indicates an improvement.
  scores on a scale at baseline | 55.01 (21.58) | 56.57 (20.61) | 55.65 (21.01)

OUTCOME MEASURES:

1. Primary Outcome: The Tinnitus Functional Index
Description: A self-reported outcome measure of tinnitus severity. Units of measurement: scores on a scale Abbreviation TFI Minimal value: 0 Maximum value 100 Higher score is a worse outcome Units are scores on a scale Total score out of 100 is reported and not any subscales Scores below 25 indicate mild tinnitus, from 25-50 indicated significant tinnitus and from 50-100 severe tinnitus
Time Frame: At baseline and at 8 weeks post-intervention
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention results: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention results | 22.85 (19.26) | 32.51 (23.28)
  Baseline results | 55.01 (21.58) | 55.26 (11.62)

2. Secondary Outcome: Tinnitus Handicap Inventory
Description: Measure of how severe the tinnitus is Units of measurement: scores on a scale Abbreviation THI Minimal value: 0 Maximum value 100 Higher score is a worse outcome Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention. Both time points are reported
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention scores: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention scores | 17.78 (14.77) | 27.11 (21.62)
  Baseline scores | 44.57 (23.40) | 47.13 (20.31)

3. Secondary Outcome: Satisfaction With Life Scale
Description: Quality of life measure Units of measurement: scores on a scale Minimal value: 5 Maximum value 35 Higher score is a better outcome
  Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention. Both scores are reported
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention socre: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention socre | 21.00 (5.05) | 20.50 (4.95)
  Baseline Score | 18.7 (5.73) | 19.48 (5.54)

4. Secondary Outcome: Cognitive Failures Questionnaire
Description: Measure of how cognitive difficulties such as concentration and memory Units of measurement: scores on a scale Minimal value: 0 Maximum value 100 Higher score is a worse outcome Units are scores on a scale Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention
Population: clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention | 30.06 (12.89) | 33.06 (19.24)
  Baseline score | 34.93 (14.38) | 39.65 (19.31)

5. Secondary Outcome: Patient Health Questionnaire
Description: Measure of signs of depressive disorders Units of measurement: scores on a scale Minimal value: 0 Maximum value 28 Higher score is a worse outcome Total score used, not sub scales
Time Frame: At baseline and at 8 weeks post-intervention
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention | 2.78 (3.02) | 4.97 (4.54)
  Baseline score | 6.5 (5.48) | 7.98 (6.05)

6. Secondary Outcome: Generalised Anxiety Disorder
Description: Measure of anxiety disorder and traits Units of measurement: scores on a scale Minimal value: 0 Maximum value 21 Higher score is a worse outcome Total score used, not sub scales
Time Frame: At baseline and at 8 weeks post-intervention. Both scores are reported
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention | 3.33 (3.21) | 3.42 (3.60)
  baseline scores | 6.43 (5.64) | 6.78 (5.54)

7. Secondary Outcome: Hyperacusis Questionnaire
Description: Measure of abnormal sound sensitivity Units of measurement: scores on a scale Minimal value: 0 Maximum value 42 Hotal score used, not sub scales
Time Frame: At baseline and at 8 weeks post-intervention. both scores are reported
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention | 12.51 (9.01) | 12.94 (7.51)
  Baseline severity | 15.65 (9.06) | 15.65 (7.42)

8. Secondary Outcome: Hearing Handicap Inventory
Description: Measure of hearing difficulties or hearing disability using a screening tool Units of measurement: scores on a scale Minimal value: 0 Maximum value 40 Higher score is a worse outcome Total score used, not sub scales
Time Frame: At baseline and at 8 weeks post-intervention
Population: Clinical population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention | 9.11 (11.59) | 12.00 (9.56)
  Baseline score | 11.74 (10.66) | 14.3 (11.58)

9. Secondary Outcome: Insomnia Severity Index
Description: Measure of sleep problems Units of measurement: scores on a scale Abbreviation ISI Minimal value: 0 Maximum value 28 Higher score is a worse outcome Total score used, not sub scales
Time Frame: Assessed at baseline and 8 weeks post-intervention. both scores are reported
Population: Clinical population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
Number analyzed (Participants) | 46 | 46
score on a scale
  8 weeks post-intervention: number analyzed (Participants) | 37 | 37
  8 weeks post-intervention | 5.69 (4.64) | 10.03 (6.88)
  Baseline score | 11.43 (6.36) | 13.65 (6.62)

ADVERSE EVENTS:
Time Frame: 8 weeks post intervention
Description: All-Cause Mortality: Deaths related to the study Serious Adverse Events: a severe increase in tinnitus distress; anxiety or depression related to the study Other Adverse Events: A severe increase in insomnia, hyperacusis or hearing handicap
Arm/Group | Experimental Group: iCBT | Face-to-face Clinical Tinnitus Care
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

LIMITATIONS AND CAVEATS:
This trial had many challenges, such as difficulty recruiting a sufficient number of participants.

The low ratio of people participating in the study in comparison with those who were invited was a potential source of bias. In addition, the nonuniform nature of the clinical care received from the various study centers may have contributed to the variability. Interpretation of the data are limited to participants with similar demographic and clinical profiles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02665975/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT02665975/ICF_001.pdf